CLINICAL TRIAL: NCT06096519
Title: Effectiveness and Implementation of Text Messaging to Improve Human Immunodeficiency Virus (HIV) Testing in Adolescents
Brief Title: Effectiveness and Implementation of Text Messaging to Improve HIV Testing in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathryn Macapagal, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00217358; 5R01MH129207 (NIH)
Record Dates: First submitted 2023-05-18; First posted 2023-10-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: Human immunodeficiency virus; Adolescents; Sexually transmitted infections; Sexual health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Information only control (Placebo Comparator): The attention matched control arm will include information based text messages about general health and sexual health topics such as human immunodeficiency virus (HIV), sexually transmitted infections (STIs), relationships, and biomedical methods of HIV prevention (e.g., Pre-exposure prophylaxis (PrEP), Post-exposure prophylaxis (PEP)). No motivational or behavioral skill based text messages aimed at increasing HIV testing or reducing HIV risk behavior will be included. All participants will receive 8-10 messages/day for 6 weeks, with a 1 week booster. Participants in the control arm will have modified access to the interactive features such as quizzes, badges, an external chatbot feature, a website with sexual health resources and a group chat feature (a group of 3-5 total participants with whom participants can discuss program content).
  Interventions: Behavioral: Information only control arm
- Information, motivation, behavioral skills treatment arm (Experimental): The active treatment arm consists of text messages with information, motivation, and behavioral skill based text messages aimed at increasing HIV testing, our primary outcome. Secondary outcomes include STI testing, PrEP uptake, condomless sex, and discussions with providers about PrEP/HIV care. Hypothesized mediators of HIV testing include testing/prevention information, motivation, and behavioral skills. All participants will receive 8-10 messages/day for 6 weeks, with a 1 week booster session following the intervention. In the active treatment arm, participants will have full access to interactive features such as quizzes, badges, an external chatbot feature, a website with sexual health resources, and a group chat feature (a group of 3-5 total participants with whom participants can discuss program content) to promote engagement and enhance learning and skills acquisition.
  Interventions: Behavioral: Information, motivation, behavioral skills treatment arm

INTERVENTIONS:
Behavioral: Information, motivation, behavioral skills treatment arm — Our intervention will be an updated version of (Guy2Guy) G2G, a 2014 text messaging-based healthy sexuality and HIV prevention program specifically for adolescent males. The treatment arm of G2G was guided by the Information-Motivation-Behavioral Skills (IMB) model and proved to be efficacious at increasing HIV testing in 13-18 year old adolescent males. In this updated version we will continue to utilize the IMB model, but modernize the content to include updated HIV prevention information (e.g., novel methods of HIV testing, PrEP, PEP) and tailor the text-message content to meet the needs of all adolescents.
  Other Names: Guy2Guy (G2G)
  Arms: Information, motivation, behavioral skills treatment arm
Behavioral: Information only control arm — This information only control arm will consist of content and text messages focused on health behavior information, including mood, sexual health, substance use, and other health behaviors. It will be identical in length to the intervention arm.
  Arms: Information only control

SUMMARY:
This study will test the effectiveness of a text message-based intervention on human immunodeficiency virus (HIV) testing behaviors among adolescent (13-18 year old). To test the effectiveness on HIV testing behaviors we will randomize participants to the treatment or an attention matched information only control arm and asses our primary effectiveness outcome of objective HIV testing (e.g., photo of test results).

DETAILED DESCRIPTION:
Adolescents (ages 13-18) are disproportionately affected by HIV, accounting for 21% of all new infections in the U.S. in 2019. Although CDC and USPTF recommend HIV screening among adolescents, testing rates are very low (<10% have ever been tested). Furthermore, in the U.S., 44% of 13-24-year-olds who are HIV-positive are unaware of their status - the highest percentage of undiagnosed infections of all age groups.

As such there is a need for interventions that aim to increase HIV testing in adolescents. This study builds upon the work of a previous text-based sexual health intervention program called G2G. The G2G pilot randomized controlled trial showed adolescents in the active treatment arm were >3x more likely to report being tested for HIV at follow-up compared to those in the control arm. Given the success of HIV testing behaviors in G2G this current study will aim to update G2G with the latest HIV prevention and testing science, tailor the intervention content so it is modern and inclusive of all adolescents, and test its effectiveness on the outcome of validated HIV testing (e.g., photo of HIV test result). We will test this in a nationwide randomized controlled trial with 360 adolescents aged 13-18.

The primary efficacy outcome measure is HIV/STI testing via self report and objective evidence (e.g., photo of their test results) at 3 month and 6 month follow up surveys. Our study hypothesizes that participants assigned to the treatment arm of the intervention will have higher odds of having received an HIV test at 3 and 6 month follow up compared to those in the control arm. Ultimately, increased HIV testing in this group will mitigate transmission rates and improve the HIV prevention and care continua in this population.

ELIGIBILITY:
Inclusion Criteria:

* Have penetrative or oral sex in their lifetime
* 13-18 years old
* reads in English at a 8th grade level
* HIV negative or unknown status
* own a cell phone with an unlimited MMS plan and plan to have the same number during the study
* can provide informed assent, as shown on a capacity to consent assessment
* live in the U.S. or territories.

Exclusion Criteria:

* Previous lifetime testing for HIV or an STI OR no testing since last sexual experience
* HIV positive
* Currently on PrEP

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HIV/STI testing | Baseline, 3-months post-intervention, 6-months post-intervention
  Participants asked to self-report their history of HIV testing; scale item (No, I have never been tested for HIV/Yes, I have been tested HIV/ I do not know or not sure)
Most recent HIV test | Baseline, 3-months post-intervention, 6-months post-intervention
  Participants asked to provide date (open-ended) and outcome of most recent HIV test (scale item: negative/positive/I did not get the result)
Objective proof of HIV testing | through study completion, an average of 9 months, 3-months post-intervention, 6-months post-intervention
  Participants are asked to upload image of proof of most recent HIV test; open-ended (upload image)

SECONDARY OUTCOMES:
Lifetime STI testing | Baseline, 3-months post-intervention, 6-months post-intervention
  Participants asked to self-report their history of STI testing; outcomes assessed via scale items (No, I have never been tested for any STI/Yes, I have been tested for at least one STI/ I do not know or not sure)
Lifetime number of sexual partners someone has had condom-less sex with | baseline, 3-months post-intervention, 6-months post-intervention
  Incidence of Condomless Sex
Ever taken PrEP | baseline, 3-months post-intervention, 6-months post-intervention
  Binary-scale item (yes/no)
Currently taking PrEP | baseline, 3-months post-intervention, 6-months post-intervention
  Binary-scale item (yes/no)
Sexual Health Communications Scale | baseline, 3-months post-intervention, 6-months post-intervention
  This is a 7-item select all that apply question which asks participants about their communicative experiences as an adolescent receiving services from medical healthcare providers, specifically around HIV testing, PrEP, STI and HIV prevention. Question adapted from the Sexual Health Communications Scale (Fisher et al., 2018). More selected options indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No